CLINICAL TRIAL: NCT02468947
Title: Finding Ideal Blood Culture Volume in NICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Bromiker, Ruben M.D, Senior Physician NICU, Shaare Zedek Medical Center
Other Study IDs: 182/14
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Ideal Sample Volume for Blood Cultures
Keywords: Neonatal sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to assess the effectivity of different sample volumes in blood cultures.

DETAILED DESCRIPTION:
The investigators intend to compare yield of 0.5ml sample x2 vs 0.25 ml samples x2 (aerobic and anaerobic media for each volume) taken from the sample taken from the same site and time.

Time to positivity will also be compared, as well as possible contamination rates.

ELIGIBILITY:
Inclusion Criteria:

* Suspected sepsis

Exclusion Criteria:

* Need for extra puncture in order to withdraw enough blood for the second set of cultures.
* Urgent need for antibiotic without time for cultures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All babies treated in the neonatology department of the institution undergoing sepsis workup
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Positive blood cultures of each group | 2 years

SECONDARY OUTCOMES:
Time to positivity for each group | 2 years
Suspected contamination rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ruben Bromiker, Jerusalem, Israel

REFERENCES:
- [Result] Yaacobi N, Bar-Meir M, Shchors I, Bromiker R. A prospective controlled trial of the optimal volume for neonatal blood cultures. Pediatr Infect Dis J. 2015 Apr;34(4):351-4. doi: 10.1097/INF.0000000000000594. PMID 25764096